CLINICAL TRIAL: NCT06711614
Title: FIRE-Diet: Food as an Intervention to Reduce the Effects of Woodsmoke Exposure on Respiratory Health
Acronym: FIRE-Diet-M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Emily Brigham, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H23-03904
Record Dates: First submitted 2024-10-18; First posted 2024-12-02 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Healthy Individuals
Keywords: Diet Intervention; EPA; DHA; Omega-3 fatty acids

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized to begin the study with the control diet (their usual diet) or the intervention diet (aimed at increasing intake of fatty fish high in omega-3 fatty acids, fruits, and vegetables) x ~4 weeks. After a washout period of at least 4 weeks the participant will complete the alternate assignment. At the end of each assignment (control or intervention diet) the participant will undergo a controlled exposure to wood smoke x 2 hours, following which lung health outcomes will be assessed as described.
Who Masked: Investigator
Masking Description: environmental engineer (administering the woodsmoke exposure) will be masked to diet assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Diet First, then Control Diet (Other): Participants will complete ~4 weeks of the Intervention Diet, followed by a washout period of at least 4 weeks, then ~4 weeks of the Control Diet. At the end of each Diet period, participants will undergo a 2 hour controlled wood smoke exposure, following which outcome measures will be assessed.
  Interventions: Other: Intervention Diet; Other: Control Diet
- Control Diet First, then Intervention Diet (Other): Participants will complete ~4 weeks of the Control Diet, followed by a washout period of at least 4 weeks, then ~4 weeks of the Intervention Diet. At the end of each Diet period, participants will undergo a 2 hour controlled wood smoke exposure, following which outcome measures will be assessed.
  Interventions: Other: Intervention Diet; Other: Control Diet

INTERVENTIONS:
Other: Intervention Diet — Designed to increase Omega-3 Fatty Acids (Eicosapentaenoic acid (EPA), Docosahexaenoic acid (DHA)), fruit, and vegetable intake, participants will receive grocery and meal deliveries for approximately 4-weeks via online ordering with dietician counselling.
Other: Control Diet — Participants will receive weekly food subsidies for their groceries for 4-weeks (~equivalent to the subsidies to provide groceries in the Intervention arm) but are free to purchase whatever they wish. The participants will continue to have dietician counseling during this time.

SUMMARY:
Research suggests that consuming more fatty fish, fruits, and vegetables could potentially shield the lungs from the negative impacts of air pollution. The research team will look at whether a dietary intervention aimed at increasing intake of these foods can protect the lungs from woodsmoke as the air pollutant and look into how this works.

DETAILED DESCRIPTION:
This study aims to recruit 48 healthy adult volunteer participants (24 male and 24 female biologic sex assigned at birth) with no known respiratory diseases (as assessed by the study physician) who will breathe in woodsmoke while they are supported to eat a diet higher in fatty fish, fruits, and vegetables (the intervention diet), or not (the control diet).

All participants will undergo a screening visit to assess eligibility for the study. Once deemed eligible, they will experience three exposure visits: one fresh air (filtered air - FA) exposure and two woodsmoke (WS) exposures. The study will span a minimum duration of 15 weeks with 10 in-person visits to the site at Vancouver General Hospital, totaling approximately 34.5 hours. During these visits, participants will complete a series of questionnaires, sample collections (blood, urine, sputum (clumps of mucus that are coughed up from the lungs)), and lung function tests, in addition to the exposures mentioned above.

Off-site commitments will require participants to follow the recommended diet assigned at the time, complete some electronic questionnaires and breathing tests at home after exposures, and complete telephone calls with the study dietician (approximately 30-minute calls, weekly).

Participants will be provided with meal and grocery deliveries to meet intake goals specified by the study or a subsidized amount of groceries per week depending on the diet intervention assigned at that time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, and specifically with no respiratory disease
* Not taking any supplements, or willing to abstain from supplement use for 4-weeks prior to study start and the whole duration of the study,
* Must currently consume, on average, less than 2 servings of fish per week and fewer than 5 servings of fruits and vegetables per day based on screening questionnaires.
* Must have a null GSTM1 genotype determined at screening.
* Must be able to provide a sufficient sputum sample during the screening visit.

Exclusion Criteria:

* Pregnant or planning to become pregnant during the study period.
* Health conditions that would pose an unacceptable risk of dietary change, or conditions that are uncontrolled based on principal investigator's judgement.
* Actively attempting to lose weight.
* Frequent wood smoke exposure (e.g. at home or employment).
* Unable to store provided meals and food safely.
* Food allergies/intolerance or food aversion preventing adherence to the intervention diet, or unwillingness/medically unable to adjust diet in line with the intervention.
* Relocation during the study period to an area which will prevent food delivery.
* History of smoking tobacco, marijuana, or and other substance or vaping within the past 6 months, or having smoked the equivalent of 0.5 pack-years ever.
* Body mass index (BMI) <18.5, as determined during the in-person screening visit.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Within-individual change in sputum neutrophil % | Across study duration, anticipated ~15 weeks.
  Within-individual change in sputum neutrophil %, compared across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in sputum neutrophil activation and function | Across study duration, anticipated ~15 weeks
  Within-individual change in sputum neutrophil activation (expression of neutrophil activation cell surface markers, release of neutrophil elastase and myeloperoxidase), and neutrophil function (phagocytosis, intracellular oxidative burst, and extracellular trap formation) across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in airway resistance | Across study duration, anticipated ~15 weeks.
  Within-individual change in airway resistance, as measured by impulse oscillometry (resonant frequency (Fres) and peripheral airway resistance (R5-R20)) across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in sputum biomarkers of inflammation | Across study duration, anticipated ~15 weeks.
  Within-individual change in sputum biomarkers of inflammation (IL-6, IL-8, and TNF-alpha in sputum as well as fractional exhaled nitric oxide) across Intervention and Control Diet periods post wood smoke exposures.

SECONDARY OUTCOMES:
Within-individual change in sputum biomarkers/arbiters of inflammation | Across study duration, anticipated ~15 weeks.
  Within-individual change in sputum biomarkers of inflammation (MCP-1, IL-4, IL-5, IL-13, protectins, maresins, resolvins) across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in upper airway (nasal) markers of neutrophil activation and function | Across study duration, anticipated ~15 weeks.
  Within-individual change in biomarkers of neutrophil activation (myeloperoxidase, neutrophil elastase in nasal epithelial lining fluid) across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in upper airway (nasal) biomarkers/arbiters of inflammation | Across study duration, anticipated ~15 weeks.
  Within-individual change in biomarkers of inflammation (including IL-6, IL-8, TNF-alpha, MCP-1, IL-4, IL-5, IL-13, protectins, resolvins, maresins in nasal epithelial lining fluid) across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in blood neutrophil % | Across study duration, anticipated ~15 weeks.
  Within-individual change in blood neutrophil %, compared across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in blood neutrophil activation and function | Across study duration, anticipated ~15 weeks
  Within-individual change in blood neutrophil activation (expression of neutrophil activation cell surface markers, release of neutrophil elastase and myeloperoxidase), and neutrophil function (phagocytosis, intracellular oxidative burst, and extracellular trap formation) across Intervention and Control Diet periods post wood smoke exposures.
Within-individual change in spirometry | Across study duration, anticipated ~15 weeks.
  Within-individual change in spirometry, as measured by (Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), and FEV1/FVC) across Intervention and Control Diet periods post wood smoke exposures.

OTHER OUTCOMES:
Within-individual change in systemic biomarkers/arbiters of inflammation and oxidative stress | Across study duration, anticipated ~15 weeks.
  Within-individual change in systemic biomarkers/arbiters of inflammation (including IL-6, IL-8, TNF-alpha, MCP-1, IL-4, IL-5, IL-13, resolvins, maresins, protectins in blood) and oxidative stress (including urinary leukotrienes) across Intervention and Control Diet periods post wood smoke exposures.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Brigham, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada